CLINICAL TRIAL: NCT00193765
Title: Elective Versus Therapeutic Neck Dissection in the Treatment of Early Node Negative Squamous Cell Carcinoma of the Oral Cavity
Brief Title: Elective vs Therapeutic Neck Dissection in Treatment of Early Node Negative Squamous Carcinoma of Oral Cavity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, A K D'Cruz, MS, DNB, FRCS (Hon.), Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH/131/2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Oral Cancer
Keywords: neck dissection; survival; early oral cancer; Early oral cavity squamous cancer with node negative neck
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait and Watch (Active Comparator): Therapeutic neck dissection on developing nodal relapse
  Interventions: Procedure: Therapeutic Neck Dissection
- Elective Neck dissection (Experimental): Elective neck dissection in early oral cancer at the time of primary surgery
  Interventions: Procedure: Elective neck dissection in early oral cancer

INTERVENTIONS:
Procedure: Elective neck dissection in early oral cancer — Elective neck dissection in early node negative oral cancers at the time of primary surgery
  Other Names: Early oral cancer; Node negative neck
  Arms: Elective Neck dissection
Procedure: Therapeutic Neck Dissection — There is no active intervention for the neck at the time of primary surgery. Therapeutic Neck Dissection at the time of nodal relapse
  Other Names: Wait & Watch
  Arms: Wait and Watch

SUMMARY:
Cervical nodal metastasis is the single most important prognostic factor in head and neck cancers. Appropriate management of the neck is therefore of paramount importance in the treatment of these cancers. While it is obvious that the positive neck must be treated, controversy has always surrounded the clinically node negative neck with respect to the ideal treatment policy.The situation is difficult with regards to early cancers of the oral cavity (T1/T2). These cancers are usually treated with surgery where excision is through the per-oral route. Elective neck dissection in such a situation is an additional surgical procedure with its associated costs, prolonged hospitalization and may be unnecessary in as high as 80% of patients who finally turn out to be pathologically node negative. Should the neck be electively treated or there be a wait and watch policy? Current practice is that the neck is always addressed whenever there is an increased propensity to cervical metastasis or when patient follow-up is unreliable.

There is clearly a need therefore for a large randomized trial that will resolve the issue either way once and for all.

Primary Objective:

To demonstrate whether elective neck dissection (END) is equal or superior to the wait and watch policy i.e.

therapeutic neck dissection (TND) in the management of the clinically No neck in early T1 /T2 cancers of the oral cavity.

Secondary Objective:

1. Does Ultrasound examination have any role in the routine initial workup of a node negative patient?
2. How are patients ideally followed up -does sonography have a role or is clinical examination sufficient.
3. Is assessment of tumor thickness by the surgeon at the time of initial surgery accurate -Is there a correlation
4. Identify histological prognostic factors in the primary that may help identify a sub-set of patients at an increased risk for cervical metastasis.

DETAILED DESCRIPTION:
Stratification criteria:

1. Size
2. Sex
3. Site
4. Sonography

Randomization (I): All patients will be randomly allocated into one of two arms: wait and watch policy group or elective neck dissection group. Both arms will have similar wide excision of primary tumor in oral cavity per oral route.

Randomization (II): Following surgery and after complete recovery prior to discharge, patients will be randomized a second time for follow-up into two arms namely clinical examination versus clinical examination and ultrasonography of neck.

SURGICAL PROCEDURE:

Primary: tumor will be excised after proper exposure via per-oral route.

* Emphasis will be to achieve a wide clearance with tumor free margins to obviate need of subsequent radiotherapy to primary, which would otherwise act as a confounding factor.

Neck: Patients randomized to neck dissection will undergo a standard supra-omohyoid neck dissection that will involve clearance of nodal Levels I, II, and III.Completion MND will be done as and when required. Patients who develop metastatic adenopathy on follow-up will undergo a modified neck dissection/radical neck dissection depending on size of metastatic disease. Those who have nodes suggestive of metastasis on follow-up sonography, will undergo a supraomohyoid dissection, frozen section followed by a modified neck dissection if positive.

Depth of tumor infiltration though probably most important individual prognostic factor in deciding likelihood of cervical metastasis, is unfortunately only available to clinician with final histopathology report. Had this parameter been present at time of surgery patient with an increased likelihood of metastasis could have undergone an elective neck dissection while those with a lower incidence could have been saved an unnecessary operation .This study would help find out accuracy of correlation between gross assessments of thickness by surgeon, on frozen section with final thickness on histopathology and would be of importance in a country like ours where oral cancers are very common and facilities of frozen as well as expertise to measure accurately tumor thickness at histopathology may be unavailable.

END POINT OF STUDY:

The primary end point will be overall survival and secondary end point will be DFS. The patients will be followed up until death or study close whichever is earlier. Since overall survival is the primary endpoint, patients will be followed up until death. telephonic or mail contact is acceptable.

Local failures, distant metastasis and second primary will be documented.

DATA COLLECTION, QUALITY CONTROL & ANALYSIS:

Assuming baseline overall survival of 60%, for expected improvement in treatment arm of 10% no. of patients required will be is 710 (355 in each arm) with α=0.05 (one sided) & power of 80% (β=20). An interim analysis is planned at 250 events (death) occur.

Ultrasound in routine follow-up of all patients will be labor intensive. However median follow-up to recurrence in all studies both retrospective/prospective has been 9 months on an average (range 6 months- 13months). It will therefore be important to follow patients every vigilantly in first 12 months from primary treatment. Follow-up schedules will be: First visit: 4 weeks;First 6 months: 4-6 weeks; 6-12 months: 6-8 weeks; 12 months- 2 years: 8-12 weekly; Thereafter: 3 monthly.

Patients will be encouraged and counseled to come for check up on earlier date within range allowed. All patients will be followed up by one of investigators and entry made both in source document as well as central registration cell at CRS with study coordinator. At each examination patients will undergo a through head and neck examination as well as an ultrasound if randomized to that arm.

SUMMARY OF PROTOCOL AMENDMENTS The first version of the protocol (hereafter called Version 1) received approval from the Institutional Ethics Committee in September 2003.The most recent version of the protocol (hereafter called Version 4) received approval from the Institutional Ethics Committee in June 2014.

Version 1 dated: September 2003 Version 2 dated: December 2008 Version 3 dated: August 2011 Version 4 dated: June 2014

The number of prospective randomized controlled trials previously reported and reviewed is three in version 1 and the number of prospective Randomized controlled trial previously reported and reviewed has increased to four in version 4. The change was done in version 3.

Pre randomization USG findings for lymph nodes were not considered for eligibility criteria. Therefore patients with normal, indeterminate and those suggestive of metastasis were eligible for trial inclusion in version 1 and Patients with pre randomization ultrasound neck findings suggestive of metastasis were excluded in version 4. The change was done in version 2.

Based on pre-randomization ultrasound neck findings, patients were stratified between those with normal versus indeterminate versus suspicious for metastasis in version 1 and Patients stratification was between normal versus indeterminate ultrasound findings in version 4. The change was done in version 2

Patients and investigators blinded to pre- randomization ultrasound neck findings in version 1 and Patients and investigators are no longer blinded to pre- randomization ultrasound neck findings in version4. The change was done in Version 2

The end points are locoregional recurrence survival in version 1 and The secondary endpoint of the study has been explicitly clarified to be disease-free survival in version 4. The change was done in Version 3.

'Nodal relapse' and 'Regional Recurrence' have been defined explicitly in version 4. The change was done in version 3.

Ethical Concerns:

Protocol amendment details:

Protocol amendment was accepted by scientific ethics committee/Instititional Review board on 29/12/2008 as follows:

All patients will undergo a pre randomization ultrasonography of neck. If USG report suggests metastasis patients would be treated according to merit to avoid ethical concerns and if USG report is normal or indeterminate, patients would be randomized for trial. This protocol amendment is done in view of following 2 reasons.

Very often patients are uncomfortable to give consent when they are explained that initial ultrasonography report will be blinded and findings will not be considered in deciding patient's treatment plan. This resulted in lower recruitment of patients and it also raised ethical issues when blind was not adequately maintained especially if sonography suggested metastasis.

To overcome a difference of opinion amongst examining clinicians about a clinically significant node.

However, breaking blind would have no bearing on outcome / impact of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven T1 or T2 N0 M0 (clinical) squamous cell carcinoma of the buccal mucosa, lower alveolus, oral tongue and floor of mouth.
2. Surgery is the preferred treatment and the primary tumor can be excised with clear margins via the per-oral route.
3. No history of a prior malignancy in the head and neck region.
4. No prior malignancy outside the head and neck region in the preceding 5 years.
5. Patient will be reliable for follow-up
6. Age> 18 years and < 75 years.
7. No significant co-morbid conditions - ASA grade II and I.
8. Understands the protocol and is able to give informed consent.

Exclusion Criteria:

1. Prior radiotherapy or surgery for malignancy in the head and neck region.
2. Non squamous cell carcinomas of the oral cavity.
3. Upper alveolus and palatal lesions where there is a possibility of retropharyngeal node involvement.
4. Per-oral excision of tumor will compromise margins in the opinion of the treating surgeon.
5. Significant co-existing pre-malignant conditions like erytho-leucoplakia and oral sub mucous fibrosis that in the opinion of the clinician would interfere in the planned treatment management of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2004-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 5 years
  survival would be calculated as time period between date of randomization and date of death from any cause or last follow up

SECONDARY OUTCOMES:
Disease free survival | 5 years
  the interval between the date of randomization and the date of the first documented evidence of relapse at any site (local, regional, metastatic, or second primary) or death from any cause, whichever came first
Role of ultrasound examination in routine initial workup of a node negative patient. | 5 years
  to see that the addition of USG to routine initial work up helps in detection of cervical metastasis better
Role of ultrasonogrphy vs clinical examination in ideal follow up of patient. | 5 years
  to see if the addition of USG to routione clinical examination helps in early detection of the cervical metastasis and hence improves survival
Correlation between the tumour thickness assessment by surgeon on table , on frozen section and final histopathology. | Within 2 weeks after surgery
  to assess the concordance between the assessment on table by surgeon, pathologist at frozen section and histopathology taking histopathology as gold standard
Identify histological prognostic factors in primary that may help identify a sub-set of patients at an increased risk of cervical metastasis. | upto 5 years
  statistical analysis to identify the factors predicting cervical metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Anil K D'cruz, MS,DNB, Principal Investigator — Tata Memorial Hospital,Mumbai,India
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Worthington HV, Bulsara VM, Glenny AM, Clarkson JE, Conway DI, Macluskey M. Interventions for the treatment of oral cavity and oropharyngeal cancers: surgical treatment. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD006205. doi: 10.1002/14651858.CD006205.pub5. PMID 37650478
- [Derived] D'Cruz AK, Vaish R, Kapre N, Dandekar M, Gupta S, Hawaldar R, Agarwal JP, Pantvaidya G, Chaukar D, Deshmukh A, Kane S, Arya S, Ghosh-Laskar S, Chaturvedi P, Pai P, Nair S, Nair D, Badwe R; Head and Neck Disease Management Group. Elective versus Therapeutic Neck Dissection in Node-Negative Oral Cancer. N Engl J Med. 2015 Aug 6;373(6):521-9. doi: 10.1056/NEJMoa1506007. Epub 2015 May 31. PMID 26027881